CLINICAL TRIAL: NCT00022295
Title: Phase IB Study of Phenoxodiol Given by Constant Intravenous Infusion in Patients With Solid Neoplasms (With the Exception of Breast Cancer) Whose Tumors Are Refractory to Standard Therapy
Brief Title: Phenoxodiol in Treating Patients With Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kazia Therapeutics Limited (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068802; NOVOGEN-NV06-0024; CCF-4269; NCI-V01-1663
Record Dates: First submitted 2001-08-10; First posted 2003-01-27 (Estimated); Last update posted 2013-03-26 (Estimated); Status verified 2007-03

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — phenoxodiol

INTERVENTIONS:
Drug: idronoxil

SUMMARY:
RATIONALE: Phenoxodiol may stop the growth of tumor cells by blocking the enzymes necessary for cancer cell growth.

PURPOSE: Phase I trial to study the effectiveness of phenoxodiol in treating patients who have refractory solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of phenoxodiol in patients with refractory solid tumors.
* Determine the steady-state pharmacokinetics of this drug in these patients.
* Determine the tumor response in patients treated with this drug.

OUTLINE: This is a multicenter, dose-escalation study.

Patients receive phenoxodiol IV continuously over days 1-7. Treatment repeats every 14 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of phenoxodiol until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed at 4 weeks.

PROJECTED ACCRUAL: Approximately 18-36 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed solid tumor

  * Refractory to standard therapy OR
  * No standard therapy exists
* No breast cancer
* No active CNS metastases

  * Known CNS metastases must be previously treated with radiotherapy or surgery and stable for at least 4 weeks prior to study

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* At least 3 months

Hematopoietic:

* Platelet count greater than 100,000/mm^3
* WBC greater than 3,000/mm^3
* Neutrophil count greater than 1,500/mm^3
* Hemoglobin greater than 10 g/dL (9 g/dL for women)

Hepatic:

* Bilirubin less than 1.2 mg/dL
* Transaminases no greater than 3 times upper limit of normal

Renal:

* Creatinine no greater than 1.4 mg/dL

Other:

* No active infection
* No contraindication to the insertion of a vascular access device
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent systemic anticancer immunotherapy

Chemotherapy:

* No concurrent systemic anticancer chemotherapy

Endocrine therapy:

* No concurrent systemic anticancer hormonal therapy except luteinizing hormone-releasing hormone agonists or antagonists

Radiotherapy:

* See Disease Characteristics
* Concurrent localized radiotherapy for control of local disease complications allowed

Surgery:

* See Disease Characteristics

Other:

* Recovered from prior antineoplastic therapy
* At least 4 weeks since prior investigational agents
* No other concurrent investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2001-08; Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Graham Kelly, PhD, Study Chair — MEI Pharma, Inc.
Locations (1):
- Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio, United States